CLINICAL TRIAL: NCT03575377
Title: Opioid Use, Storage, and Disposal Among Pediatric Patients After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Jennifer Cooper, Principal Investigator, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB18-00157
Record Dates: First submitted 2018-06-19; First posted 2018-07-02 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Tonsillitis; Sleep Disordered Breathing; Hernia; Hydrocele; Hypospadias; Undescended Testicle; Circumcision
MeSH Terms: conditions — Tonsillitis; Sleep Apnea Syndromes; Hernia; Testicular Hydrocele; Hypospadias; Cryptorchidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deterra Bag (Experimental): These families will receive a Deterra® bag (a drug Disposal Aid) and instructions on its use by a research team member.
  Interventions: Other: Disposal Aid
- Control (No Intervention): These families will receive routine postoperative instructions only.

INTERVENTIONS:
Other: Disposal Aid — Deterra® drug deactivation system
  Arms: Deterra Bag

SUMMARY:
Opioids are an important component of post-operative pain management among children, but are often prescribed in excess and rarely disposed of appropriately. The lack of prompt and proper opioid disposal after recovery from surgery is contributing to the opioid crisis in Ohio by placing children at risk of accidental ingestion of opioids remaining in the home and allowing for unused opioids to be diverted for non-medical use. The investigators propose to reduce the burden of the opioid crisis in Ohio by testing a strategy to increase proper opioid disposal by families of children undergoing outpatient surgery. The investigators will test the impact of a novel opioid disposal mechanism, the Deterra® drug deactivation system, after pediatric surgical operations. This system deactivates pills, liquids, or patches, allowing for their disposal in the home garbage. The investigators propose to evaluate the effectiveness of providing Deterra® bags to families of children having surgery on their disposal of excess opioids. The investigators will perform a randomized controlled trial (RCT) to test the effectiveness of Deterra® to improve opioid disposal among families of children having outpatient surgery at Nationwide Children's Hospital.

DETAILED DESCRIPTION:
Opioids are an important component of post-operative pain management among children, but are often prescribed in excess and rarely disposed of appropriately. The lack of prompt and proper opioid disposal after recovery from surgery is contributing to the opioid crisis in Ohio by placing children at risk of accidental ingestion of opioids remaining in the home and allowing for unused opioids to be diverted for non-medical use. The investigators propose to reduce the burden of the opioid crisis in Ohio by testing a strategy to increase proper opioid disposal by families of children undergoing outpatient surgery. The investigators will test the impact of a novel opioid disposal mechanism, the Deterra® drug deactivation system, after pediatric surgical operations. This system deactivates pills, liquids, or patches, allowing for their disposal in the home garbage. The investigators propose to evaluate the effectiveness of Deterra® for opioid disposal among families of Ohio children having surgery. The investigators will perform a randomized controlled trial (RCT) to test the effectiveness of Deterra® to improve proper opioid disposal among families of children having outpatient surgery at Nationwide Children's Hospital.

The goal of this project is to evaluate the impact of providing the Deterra® drug deactivation system on the excess opioid disposal rate among families of children having outpatient otolaryngologic or urologic surgery at NCH. A second objective of this study is to evaluate whether the impact of the Deterra® drug deactivation system varies by parent/guardian health literacy level or signing of an "opioid consent form" acknowledging that they will follow appropriate dosing recommendations, not give opioids if their child appears sleepy, not give Tylenol concurrently with Tylenol-containing opioid medications, dispose of unused opioids safely and responsibly, and contact their child's surgeon's office or the on-call physician with any questions. To accomplish these objectives, the investigators will perform a randomized controlled trial comparing groups of patients who receive either 1) a Deterra® bag along with brief instruction on how and why to use it along with routine postoperative instructions or 2) routine postoperative instructions.

The investigators plan to enroll 202 caregivers of children having outpatient surgery. All families will receive a 1-page pain journal to record the child's opioid and non-opioid adjunct pain medication administration. In addition to the instructions provided by the care team as described above, families randomized to the intervention arm will additionally receive a Deterra® bag and instructions on its use by a research team member.

In order to minimize disruption to the clinical work flow, minimal data will be collected at baseline directly from enrolled families. This will include the contact information required for follow-up, a limited set of research related questions, and a brief assessment of parent/guardian health literacy. Baseline demographic and clinical characteristics of the child, such as their primary payer, residential address, age, and comorbidities at the time of surgery will be extracted from the electronic medical record.

Parents/guardians will be contacted by their preferred method of email survey or phone call at 2 weeks postoperatively, at which time they will be surveyed on their child's postoperative opioid and non-opioid medication use, opioid storage location, quantity of opioid remaining, disposal method, and any barriers to disposal. If the child continues to require opioids, they will be contacted again at 4 weeks postoperatively. If the parent believes that their older child or adolescent can assist in answering the survey questions, they will be encouraged to complete the survey together. The primary outcome of this trial is the proper disposal of unused opioids. Secondary outcomes include the quantities of opioid used and leftover after surgery, opioid storage location, disposal by any method, and barriers to disposal.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian of a child having outpatient otolaryngologic or urologic surgery at Nationwide Children's Hospital
* Child's age is between 1 and 17 years
* Child is expected to receive a discharge opioid prescription

Exclusion Criteria:

•Unable or unwilling to track pain medication use or complete a follow-up survey

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 202 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Proper disposal of unused opioids | 2-4 weeks
  The proper disposal of unused opioids, defined as the disposal of unused opioids by an FDA-recommended method or by using the Deterra® drug deactivation system.

SECONDARY OUTCOMES:
Quantity of opioid used after surgery | 2-4 weeks
  Number of doses of opioid pain medication used after surgery
Quantity of opioid leftover after surgery | 2-4 weeks
  Number of doses of opioid pain medication leftover after surgery
Proper storage of opioids | 2-4 weeks
  Whether the opioids were properly stored after surgery
Barriers to opioid disposal | 2-4 weeks
  What the parent/caregiver perceived as barriers to their disposal of their child's opioids after surgery
Disposal of unused opioids by any method | 2-4 weeks
  Disposal of unused opioids by any recommended or non-recommended method

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Cooper, PhD, Principal Investigator — Research Institute at Nationwide Children's Hospital
Locations (1):
- Jennifer Cooper, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lawrence AE, Carsel AJ, Leonhart KL, Richards HW, Harbaugh CM, Waljee JF, McLeod DJ, Walz PC, Minneci PC, Deans KJ, Cooper JN. Effect of Drug Disposal Bag Provision on Proper Disposal of Unused Opioids by Families of Pediatric Surgical Patients: A Randomized Clinical Trial. JAMA Pediatr. 2019 Aug 1;173(8):e191695. doi: 10.1001/jamapediatrics.2019.1695. Epub 2019 Aug 5. PMID 31233129